CLINICAL TRIAL: NCT03032042
Title: Intestinal Microbiome Post-Azythromycin/Albendazole Treatment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We were not able to secure IRB approval in the timeline necessary to do this study.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 17-0101
Record Dates: First submitted 2017-01-08; First posted 2017-01-26 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Helminth Infection
Keywords: intestinal microbiome; soil-transmitted helminths; mass drug administration
MeSH Terms: conditions — Trematode Infections | interventions — Azithromycin; Albendazole; Treatment Delay

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- albendazole at day 0, azithromycin at day 7 (Experimental)
  Interventions: Drug: Albendazole
- azithromycin at day 0, albendazole at day 7 (Experimental)
  Interventions: Drug: Azithromycin
- albendazole at day 0, azithromycin at day 0 (Experimental)
  Interventions: Drug: Azithromycin; Drug: Albendazole
- Delayed treatment (Other): albendazole at day 7, azithromycin at day 7
  Interventions: Drug: Delayed treatment

INTERVENTIONS:
Drug: Azithromycin
  Arms: albendazole at day 0, azithromycin at day 0; azithromycin at day 0, albendazole at day 7
Drug: Albendazole
  Arms: albendazole at day 0, azithromycin at day 0; albendazole at day 0, azithromycin at day 7
Drug: Delayed treatment — Albendazole+Azithromycin
  Arms: Delayed treatment

SUMMARY:
Molecular testing of the gut microbiome and enteric pathogens is rapidly moving beyond targeted PCR testing to next generation sequencing techniques. In addition, the current state of monitoring for soil-transmitted helminth infections is moving increasingly from microscopic techniques to molecular techniques. The targeted PCR test for soil transmitted helminth diagnosis has been validated on stool samples, but not rectal swabs. Bulk stool samples are logistically challenging and time-intensive to collect, thus participation is often far from optimal. Rectal swabs are more efficient and may result in higher participation. In this study, children will be randomized to either albendazole, azithromycin, or both drugs, after which both rectal swabs and bulk stool samples will be collected. The investigators will compare the PCR test for soil transmitted helminth infections using both the rectal swabs and the bulk stool samples. In addition, the investigators will analyze the gut microbiome of the children using next generation sequencing techniques to gain insight into effects of mass drug administration.

ELIGIBILITY:
Inclusion Criteria:

* all children 0 to 5 (up to 6th birthday)

Exclusion Criteria:

* individuals with a macrolide allergy
* refusal of parent/guardian

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Microbial diversity in the intestinal microbiomes of children aged 1-60 months | Day 7
  Microbiota diversity in the intestinal microbiomes of children aged 1-60 months in azithromycin-treated, albendazole-treated, azithromycin+albendazole-treated and delayed treatment arms using phylogenetic distance measures

SECONDARY OUTCOMES:
Sensitivity of Soil-transmitted helminth infection detection in rectal swab versus bulk stool sample in children 0-5 | Day 7
  The investigators use PCR to identify soil transmitted helming infections in rectal swab samples and bulk stool sample from the same child. Using the bulk stool sample as the gold standard, the investigators will calculate the sensitivity, specificity, PPV, and NPV of the rectal swabs for detecting the various helminth infections.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Keenan, MD, MPH, Principal Investigator — F.I. Proctor Foundation, University of California San Francisco
Locations (1):
- The Carter Center Ethiopia, Addis Ababa, Ethiopia